CLINICAL TRIAL: NCT04032080
Title: Pilot Clinical Trial of Treatment With LY3023414 and Prexasertib to Inhibit Homologous Recombination (HR) in Patients With Chemotherapy-Pretreated Metastatic Triple Negative Breast Cancer (Amendment 1)
Brief Title: LY3023414 and Prexasertib in Metastatic Triple-negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 018-745
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with metastatic TNBC who meet the enrollment criteria will receive LY3023414 and prexasertib until disease progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3023414 + prexasertib (Experimental): Patients with metastatic TNBC who meet the enrollment criteria will receive LY3023414 and prexasertib until disease progression. Patients whose disease does not respond to the combination of LY3023414 and prexasertib may be treated with standard of care breast cancer therapies off study, at the recommendation of the treating physician.
  Interventions: Combination Product: Drug 1: LY3023414; Drug 2: Prexasertib

INTERVENTIONS:
Combination Product: Drug 1: LY3023414; Drug 2: Prexasertib — Metastatic TNBC patients will consent to and undergo core needle biopsies of a metastatic lesion for NGS, RPPA, and other molecular analyses at study entry.
  Patients will then be treated with 150 mg LY3023414 PO BID and prexasertib 80 mg/m^2 IV administered every 2 weeks until disease progression or unacceptable toxicity. Any time after the completion of Cycle 2 of the treatment combination, or at the physician's discretion, a second core needle biopsy of the same metastatic lesion (or different metastases if the initial metastasis has regressed) will be performed for RPPA and other molecular analyses. If a research biopsy from a patient's metastatic disease cannot be safely obtained, a skin biopsy is permitted.
  Treatment will be discontinued in patients who achieve a confirmed clinical complete response, and these patients will be followed to document the durability of the complete responses.

SUMMARY:
This study evaluates efficacy of LY3023414 and prexasertib in patients with metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
Seventy to eighty percent of breast cancers have a gene expression profile which is characterized by homologous recombination deficiency (HRD) and high proliferation. HRD leads to errors in DNA pathway [non -homologous end joining (NHEJ)] that repair DNA-breaks, a process required for metastatic triple negative breast cancer (TNBC) survival. The hypothesis of this pilot trial is that administration of LY3023414 and prexasertib will inhibit NHEJ in metastatic TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age. Patients must agree to use one highly effective (less than 1% failure rate) method of contraception or use a combination of two effective methods of contraception during treatment with study drug and for at least 12 weeks following the last dose of study drug.
2. Have a diagnosis of metastatic TNBC previously treated with standard anthracycline, cyclophosphamide, and taxane chemotherapy, unless there was a contraindication to doxorubicin, in which case prior treatment with this agent is not required. NOTE: TNBC defined as ER-negative tumors with ≤10% tumor nuclei immunoreactivity, or "ER Low Positive" as defined by the updated ASCO/CAP guidelines 2020.
3. Have not received more than 3 prior chemotherapy regimens for metastatic disease. Prior platinum and/or taxane therapy in the adjuvant or metastatic setting is permitted.
4. Have locoregional (eg, breast, chest wall, regional lymphatic) or pulmonary or hepatic metastatic disease that is amenable to core needle biopsy. If a research biopsy from a patient's metastatic disease cannot be safely obtained, a skin biopsy is permitted. If a skin biopsy cannot be safely obtained, patients may still be eligible, per physician discretion.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
6. Have adequate hematologic function, defined by:

   1. Absolute neutrophil count (ANC) >1500/mm^3
   2. Platelet count ≥100,000/mm^3
   3. Hemoglobin ≥9 g/dL
7. Have adequate liver function, defined by:

   1. AST and ALT ≤2.5 x the upper limit of normal (ULN) or ≤5 x ULN in presence of liver metastases
   2. Total bilirubin ≤1.5 x ULN
8. Have adequate renal function, defined by:

   a. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance of ≥60 ml/min
9. Have the ability to swallow oral medications
10. Patients who have a history of brain metastasis are eligible for the study provided that all the following criteria are met:

    1. Brain metastases which have been treated
    2. Off-treatment with steroids for 2 weeks before administration of the first dose of LY3023414 and prexasertib
    3. No ongoing requirement for dexamethasone or anti-epileptic drugs
    4. No clinical or radiological evidence of progression of brain metastases
11. Patient must be accessible for treatment and follow-up.
12. All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Have a family history of long QT Syndrome and serious cardiac conditions.
2. Have QTcF interval of >470 msec on screening electrocardiogram (ECG) as well as on pre-dose Cycle 1 Day 1 ECG
3. Have insulin-dependent diabetes mellitus. Patients with a type 2 diabetes mellitus are eligible if adequate control of blood glucose level is obtained by oral anti-diabetics as documented by HbA1c <8%. Patients with type 1 diabetes mellitus are not eligible.
4. Previous radiotherapy for metastatic disease completed <2 weeks prior to study treatment initiation.
5. Women who are pregnant or lactating.
6. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as:

   1. severe impaired lung functions as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
   2. liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
   3. viral hepatitis or HIV.
7. Concurrent use of CYP3A4 inhibitors and inducers from 72 hours prior to initiation of study treatment until the end of treatment.
8. History of any other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug, or that might affect interpretation of the results of this study, or render the patient at high risk for treatment complications.
9. Patients who have received prior PI3K or CHK therapy.
10. Any other investigational or anti-cancer treatments while participating in this study
11. Any other active malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A O'Shaughnessy, MD, Principal Investigator — Baylor Scott and White University Medical Center
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LY3023414 + Prexasertib: Patients with metastatic TNBC who meet the enrollment criteria will receive LY3023414 and prexasertib until disease progression. Patients whose disease does not respond to the combination of LY3023414 and prexasertib may be treated with standard of care breast cancer therapies off study, at the recommendation of the treating physician.
  Drug 1: LY3023414; Drug 2: Prexasertib Patients will be treated with 150 mg LY3023414 PO BID and prexasertib 80 mg/m^2 IV administered every 2 weeks until disease progression or unacceptable toxicity. Treatment will be discontinued in patients who achieve a confirmed clinical complete response, and these patients will be followed to document the durability of the complete responses.
Period: Overall Study
Arm/Group | LY3023414 + Prexasertib
Started | 10
Completed | 4
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | LY3023414 + Prexasertib
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 57.5 [43 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Primary Tumor Size [Mean (Standard Deviation); unit: mm] | 14.5 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy (Objective Response Rate)
Description: To assess the objective response rate associated with LY3023414 and prexasertib in metastatic TNBC patients. Objective response is measured as prolonged clinical benefit; clinical benefit is defined as progression free survival on study therapy for at least 6 months.
Time Frame: Through study completion, approximately 2 years and 8 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | LY3023414 + Prexasertib
Number analyzed (Participants) | 10
Participants | 3

2. Secondary Outcome: Efficacy (Duration of Response)
Description: To assess duration of response to combination of LY3023414 and prexasertib in metastatic TNBC patients. Duration of response is measured as prolonged clinical benefit; clinical benefit is defined as progression free survival on study therapy for at least 6 months.
Time Frame: From the time that 6 months of progression free survival on study therapy was first met until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year.
Population: All participants who received at least one dose of treatment.
Measure: Median (Full Range); unit: weeks
Arm/Group | LY3023414 + Prexasertib
Number analyzed (Participants) | 10
weeks | 9 [1 to 45]

ADVERSE EVENTS:
Time Frame: For up to 30 days following last treatment dose, approximately 7 months
Description: All AEs are assessed and recorded during treatment and for up to 30 days following the last dose of study treatment, approximately 7 months.
Arm/Group | LY3023414 + Prexasertib
All-Cause Mortality (participants affected / at risk) | 8/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3023414 + Prexasertib (N=10)
Neutrophil count decrease (Investigations) | 1 (1) — resulted in neutropenic sepsis
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3023414 + Prexasertib (N=10)
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Abnormal HBA1C (Investigations) | 2 (2)
Abnormal LVEF (Cardiac disorders) | 1 (1)
Axillary Cellulitis (Infections and infestations) | 1 (1)
Axillary Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Axillary Swelling (Blood and lymphatic system disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Chest Pressure (General disorders) | 1 (1)
Chills (General disorders) | 2 (3)
Cognitive Changes (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (15)
Dry Mouth (General disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphagia (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (3)
Encephalopathy (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 8 (8)
Fever (General disorders) | 2 (3)
Gastroesophageal Reflux Disease (GERD) (Gastrointestinal disorders) | 3 (3)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (8)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Investigations) | 1 (2)
Influenza (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Muscle Pain - Upper Limb (Musculoskeletal and connective tissue disorders) | 2 (3)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Cramping (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) — resulted in loose eyelashes
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Macular Edema (Eye disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (11)
Neutrophil Count Decreased (Investigations) | 4 (6)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Chest Wall Redness (Skin and subcutaneous tissue disorders) | 1 (1)
Localized Edema (General disorders) | 1 (1) — Edema of the neck
Paresthesia (Nervous system disorders) | 1 (1) — Right side numbness
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Right Clavicular Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 6 (6) — Stomatitis
Edema Limbs (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 6 (12)
Thrombocytosis (Investigations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Edema Cerebral (Nervous system disorders) | 1 (1) — Vasogenic Cerebral Edema
Visual Disturbances (Eye disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (9)
Weight Loss (Investigations) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 2 (4) — Worsening Anemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT04032080/Prot_SAP_000.pdf